CLINICAL TRIAL: NCT07169955
Title: The Effect of Motivational Interviewing on Low Back Pain-Related Disability Level and Quality of Life in Patients With Lumbar Discectomy
Brief Title: The Effect of Motivational Interviewing on Patients With Lumbar Discectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Keziban OZTURK, Research assisstant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-1170
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lumbar Disc Surgery; Motivational Interviewing; Nursing Care
Keywords: motivational interviewing; lumbar discectomy; nursing care; oswetry low back pain disability; quality of life
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational İnterviewing Group (Experimental): patients who underwent lumbar discectomy surgery for the first time and whose discharge was planned, not having any complications before and after disc surgery (fecal and urinary incontinence, foot drop, cauda equina syndrome, tingling, numbness, etc.), being 18 years of age or older, having no spine or musculoskeletal problems other than disc herniation.
  Interventions: Other: Motivational Interviewing
- Control Group (No Intervention): patients who underwent lumbar discectomy surgery for the first time and whose discharge was planned, not having any complications before and after disc surgery (fecal and urinary incontinence, foot drop, cauda equina syndrome, tingling, numbness, etc.), being 18 years of age or older, having no spine or musculoskeletal problems other than disc herniation,

INTERVENTIONS:
Other: Motivational Interviewing — Implementation of the Research in the Experimental Group Since the patients in the experimental group come from many different cities and regions, the interviews will be conducted online. It was planned to conduct weekly online individual motivational interviews with the patients for 40 minutes on one day of the week for 6 weeks. In the last session of the motivational interview (6th week), Oswetry Low Back Pain Disability Index and World Health Organization Quality of Life Scale - Short Form will be administered. Post-tests will be administered 6 weeks after these forms are administered. Three months (12 weeks) after the first interview, the tests will be administered again.
  Arms: Motivational İnterviewing Group

SUMMARY:
Abstract Objective: The aim of the study was to determine the effect of motivational interviewing about adaptation to body mechanics on the level of disability due to low back pain and quality of life in patients with lumbar discectomy surgery.

Method: The design of the study was a randomized controlled clinical trial with a pretest-posttest and follow-up design with a control group. The study will be conducted with patients who are hospitalized in the neurosurgery clinic of a university hospital, who have undergone discectomy surgery and whose discharge is planned. The data will be collected using the Participant Information Form, the Scale for Assessing Adaptation to Body Mechanics for Individuals with Lumbar Disc Herniation, the Motivational Interviewing Change Cycle Determination Form, the Oswetry Low Back Pain Disability Index and the World Health Organization Quality of Life Scale-Short Form. Motivational interview was applied to the experimental group. Motivational interviewing will be conducted for 6 sessions.

DETAILED DESCRIPTION:
Research Aim This research aims to contribute to the empowerment of patients in their home care processes following discectomy surgery; to enable them to perform daily living activities by moving in accordance with body mechanics and to motivate them in this regard; to reduce limitations in daily life caused by back pain; and to improve quality of life.

Research Hypotheses H1-0: There is no difference in the level of disability caused by back pain between lumbar discectomy patients who underwent MG related to adaptation to post-discharge body mechanics and those who did not.

H1: There is a difference in the level of disability caused by back pain between lumbar discectomy patients who underwent MG related to adaptation to post-discharge body mechanics and those who did not.

H2-0: There is no difference in quality of life between lumbar discectomy patients who underwent MG related to adaptation to body mechanics after discharge and those who did not.

H2: There is a difference in quality of life between lumbar discectomy patients who underwent MG related to adaptation to body mechanics after discharge and those who did not.

METHOD Study Design The study design is a randomized controlled clinical trial with pre-test, post-test, and follow-up designs and control groups.

Study Sample and Setting The study will be conducted with patients hospitalized in the neurosurgery clinic of a university hospital in Turkey who have undergone discectomy surgery and are scheduled for discharge. Power analysis was used to calculate the study sample. The sample size was calculated using the (G*PowerVersion 3.1.9.2) software package based on the study by Reyes and Aguilera (16). The number of patients planned to be included in the study was determined to be 60, with 30 patients in each group, assuming a 5% margin of error, 85% power, and an effect size of 0.79. According to the literature, the dropout rate during the research process was predicted to be 20%, so the study was planned to include 36 patients in each group.

Randomization and Group Assignment Patients will be randomly assigned to experimental and control groups to reduce bias in the study and control variables that may affect outcome parameters. The stratified block randomization method will be applied in the study, and randomization is planned to be performed by a statistician other than the researchers. In experimental studies, it is desired that the number of patients in the groups be equal or balanced, and that they also be similar regarding prognostic factors (diagnosis, age, gender, etc.). In the study, to ensure the homogeneity of each group, the motivational interviewing change phase (pre-contemplation, contemplation) will be accepted as a stratum, and a randomization list consisting of 2 stratified blocks will be created using the stratified block randomization method.

To minimize bias in the study, an independent statistician will generate a set of numbers for the intervention and control groups from strata determined using the www.randomizer.org computer software program. A randomization list will be created by randomly assigning participants to the experimental and control groups. During the assignment, the intervention and control groups will be coded as "1" and "2." Using the coin toss method, the researcher will determine which of the numbers "1" and "2" will be the experimental or control group. Sealed opaque envelopes prepared by the independent statistician according to the 4-block randomization list will be given to the researcher. The research report will be prepared according to the CONSORT 2025 guidelines.

Blinding Participants and those conducting the study will not know who is in the experimental and control groups until the study begins; a blinded technique will be applied. Due to the nature of the study, it is impossible to blind the researcher administering the intervention or the participant; however, the statistical analysis and report writing process will be blinded. Patients in the experimental and control groups will be informed about the purpose of the study. The researcher will know which participants are in the experimental group and which are in the control group. For this reason, neither single nor double blinding will be possible in this study. The data will be coded as "A" and "B" without specifying the experimental and control groups. A statistician will analyze the data coded by the group. After the statistical analyses are performed and the research report is written, the coding for the experimental and control groups will be disclosed. This blinding technique will control for selection, assignment, statistical, and reporting biases.

Data Collection Tools Data will be collected using the Body Mechanics Adaptation Assessment Scale for Individuals with Lumbar Disc Herniation, the Motivational Interviewing Change Cycle Identification Form, the Participant Information Form, the Oswetry Back Pain Disability Index, and the World Health Organization Quality of Life Questionnaire-Short Form.

Pre-Implementation After obtaining research permits, a pre-implementation will be conducted on 10% of the sample size (a total of 8 patients, four from each group) who underwent discectomy surgery at the neurosurgery clinic and met the inclusion criteria for sampling. This is to determine the feasibility of the data collection forms and the study's implementation method. After the pre-application, necessary corrections will be made to the data collection forms and the implementation of the study. Patients included in the pre-application will not be included in the sample group.

Application Patients diagnosed with lumbar disc herniation at the Brain and Nervous System Surgery Clinic and scheduled for discectomy surgery will be informed about the purpose and application of the study during the preoperative period. After obtaining patient consent, the Body Mechanics Compliance Assessment Scale for individuals with lumbar disc herniation will be administered. The study will include patients based on the value obtained in this form. The motivational interviewing change cycle identification form will be administered to patients who meet the specified criteria. The motivational interviewing change cycle form will determine the patients' place in the change cycle. After this stage, the study group will include those in the pre-contemplation and contemplation stages. The Participant Information Form, Oswetry Low Back Pain Disability Index, and World Health Organization Quality of Life Questionnaire-Short Form will be administered to patients included in the study group. Patients included in the study in the postoperative period will be interviewed again. The Oswetry Low Back Pain Disability Index and the World Health Organization Quality of Life Scale-Short Form will be administered. An appointment date will be set for a motivational interview. Subsequently, patients will be assigned to groups according to the randomization list. Motivational interviews are planned to be conducted one week after discharge.

Data Analysis The statistical evaluation of the data obtained in the study will be performed using the SPSS program. In the evaluation of the data, descriptive statistics such as frequency, percentage, arithmetic mean (X̅), and standard deviation (SD) will be used to analyze sociodemographic characteristics. The Kolmogorov-Smirnov or Shapiro-Wilk test statistic will be used to assess the normality of the data distribution. The relationship between the scales will be assessed using the correlation coefficient. Additionally, the effect size will be calculated in the study. Cronbach's Alpha coefficient will be used to assess the reliability of the scales. In the study, an Intention to Treat (ITT) analysis is planned to maintain randomization and prevent bias in case of participant dropout. The data in the study will be analyzed at a significance level of p< .05 with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* being in the pre-intention or intention stage according to the motivational interviewing change cycle determination form,
* low and medium scores on the body mechanics adaptation assessment scale for individuals with lumbar disc herniation, patients who underwent lumbar discectomy surgery for the first time and whose discharge was planned,
* The exclusion criteria were not having any complications before and after disc surgery (fecal and urinary incontinence, foot drop, cauda equina syndrome, tingling, numbness, etc.),
* volunteering to participate in the study, having no problems in speaking and understanding Turkish, being 18 years of age or older,
* having no spine or musculoskeletal problems other than disc herniation,
* having a smartphone and internet access.

Exclusion Criteria:

* having a psychiatric diagnosis,
* being in the preparation, action or maintenance phase of change,
* planning to participate in any rehabilitation program for the first 12 weeks after surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2026-01-29 (Actual)

PRIMARY OUTCOMES:
Oswetry Low Back Pain Disability Index | At 6 weeks after discharge
  The scale defined by Fairbanks (1980) and later modified by Hudson Cook (2004) is recommended as a sensitive scale for measuring functional disability in patients with low back pain due to its validity and reliability. Turkish validity and reliability was performed by Yakut et al. (2004). The Cronbach's alpha value of the scale was found to be 0.918 at day 1 and 0.895 at day 7 (Yakut et al., 2004). The form includes 10 questions, each question has 6 options ranging from 0 to 5 points. The patient is asked to choose the statement that best describes his/her condition. The highest score obtained from the scale is 50, and 1-10 points are considered as mild functional disability, 11-30 points as moderate functional disability, and 31-50 points as severe functional disability
World Health Organization Quality of Life Scale-Short Form | At 6 weeks after discharge
  It is an international quality of life assessment scale developed by WHOQOL-BREF. It consists of a total of 26 questions assessing four domains: physical, mental, social and environmental. The WHOQOL-BREFTR version consists of 27 questions with one national question added during Turkish validity and reliability studies. The questions were asked to be answered considering the last 15 days.

SECONDARY OUTCOMES:
Oswetry Low Back Pain Disability Index | At 12 weeks after discharge
  The scale defined by Fairbanks (1980) and later modified by Hudson Cook (2004) is recommended as a sensitive scale for measuring functional disability in patients with low back pain due to its validity and reliability. Turkish validity and reliability was performed by Yakut et al. (2004). The Cronbach's alpha value of the scale was found to be 0.918 at day 1 and 0.895 at day 7 (Yakut et al., 2004). The form includes 10 questions, each question has 6 options ranging from 0 to 5 points. The patient is asked to choose the statement that best describes his/her condition. The highest score obtained from the scale is 50, and 1-10 points are considered as mild functional disability, 11-30 points as moderate functional disability, and 31-50 points as severe functional disability
World Health Organization Quality of Life Scale-Short Form | At 12 weeks after discharge
  It is an international quality of life assessment scale developed by WHOQOL-BREF. It consists of a total of 26 questions assessing four domains: physical, mental, social and environmental. The WHOQOL-BREFTR version consists of 27 questions with one national question added during Turkish validity and reliability studies. The questions were asked to be answered considering the last 15 days.

CONTACTS AND LOCATIONS:
Overall Officials: Keziban Öztürk, MSc, Principal Investigator — Gazi University
Locations (1):
- Gazi Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This research is a doctoral thesis. Therefore, it is not possible to share the relevant dataset until the thesis is complete and its manuscript wil be published.